CLINICAL TRIAL: NCT00442884
Title: Effect of Acute Psychological Stress on Glucose Concentrations in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: EK-1261
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2007-03-05 (Estimated); Status verified 2007-03

CONDITIONS: Type 2 Diabetes
Keywords: glucose control in acute stress
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Psychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Trier Social Stress Test (TSST)

SUMMARY:
The study is designed to evaluate the effects of acute psychological stress on blood glucose levels. We will study one group of patients in the fasting state on a control day and a stress test day, another group will undergo the same protocol in the postprandial state.

DETAILED DESCRIPTION:
Patients with type 2 diabetes often complain about changing blood glucose levels in times of emotional or mental stress, most subject's self-reporting higher blood glucose measurements in stressful conditions. To daily distress in diabetes additional emotional or mental stress can add a further momentum to destabilize glucose levels due to the adrenocortical response with enhancing insulin resistance and decreasing the endogenous insulin secretion. Another physiological link between stress and diabetes might be a higher sensitivity of the hypothalamo-pituitary-adrenal axis, leading to antagonizing effects on insulin actions. A study in type 2 diabetes demonstrated that stressors can destabilize blood glucose levels. Stress levels in diabetes have been shown to have a relationship to diabetic complications. Previous studies of psychological stress in type 1 diabetes have shown no effect of elevated catecholamine levels after short-lived psychological stimuli on glucose levels, but a significantly delayed decrease of glucose concentrations after an acute psychological stress in the postprandial state in association with elevated cortisol levels, showing no change of glucose concentration in the fasting state. This was in contrast to previous data in healthy subjects, showing that low glucose levels before a psychological stress prevented the stress-induced activation of the hypothalamus pituitary adrenal axis, but postprandial higher blood glucose levels induced a large cortisol response. These findings of a different cortisol responses in the fasting or fed status in healthy or absolute insulin deficient subjects could also be relevant for glucose metabolism in subjects with type 2 diabetes.

The effect of an acute psychological stress on glucose concentration may critically depend on whether stress is applied in the fasting or fed state. A different metabolic response to stress depending on food intake could explain different findings in other clinical trials and contribute to understanding glucose responses to stress. The aim of our study was thus to test whether the effect of acute psychological stress on glucose concentrations is different in the fasting compared to the fed state in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* oral antidiabetic treatment and/or long acting insulin overnight

Exclusion Criteria:

* full insulin regimen
* pregnancy or breast-feeding
* instable coronary heart disease
* poor visibility
* proliferative diabetic retinopathy
* uncontrolled arterial hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-02; Study Completion 2006-08

PRIMARY OUTCOMES:
change of glucose measurements after stress test in the fasting and fed state

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wiesli, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital of Zurich, Division of Endocrinology and Diabetes, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Faulenbach M, Uthoff H, Schwegler K, Spinas GA, Schmid C, Wiesli P. Effect of psychological stress on glucose control in patients with Type 2 diabetes. Diabet Med. 2012 Jan;29(1):128-31. doi: 10.1111/j.1464-5491.2011.03431.x. PMID 21883440